CLINICAL TRIAL: NCT07072273
Title: Open-label Clinical Trial Evaluating an Emollient With Lactobacillus Reuteri for the Treatment of Pediatric Atopic Dermatitis
Brief Title: A Clinical Trial Evaluating a Probiotic Emollient for the Treatment of Pediatric Atopic Dermatitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Biogaia New Sciences AB (Industry)
Collaborators: Bioithas SL (Industry)
Responsible Party: Sponsor
Organization: BioGaia AB (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BNS_RD_002
Record Dates: First submitted 2025-07-09; First posted 2025-07-18 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Atopic Dermatitis
Keywords: AD; Atopic Dermatitis; probiotic; Eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Probiotic Ointment (Experimental): Twice-daily application for 8 weeks of an emollient topical formulation containing Lactobacillus reuteri
  Interventions: Other: Probiotic Ointment

INTERVENTIONS:
Other: Probiotic Ointment — Ointment containing Lactobacillus reuteri

SUMMARY:
The goal of this study is to evaluate the efficacy of the emollient topical formulation containing Lactobacillus reuteri in improving atopic dermatitis symptoms in children.

ELIGIBILITY:
Inclusion Criteria:

Pediatric patients of both sexes, aged between 6 months and 12 years, with a confirmed diagnosis of AD based on Hanifin and Rajka criteria (ANNEX VIII).

SCORAD index between 20 and 50, inclusive.

Signed informed consent by parents or legal guardians.

Exclusion Criteria:

History of phototherapy for the treatment of AD.

Previous treatment with biologic agents or JAK inhibitors for AD.

Use of systemic corticosteroids within one month prior to inclusion in the clinical trial.

Use of topical corticosteroids within one month prior to inclusion in the clinical trial.

Use of conventional systemic immunosuppressants for AD (e.g., azathioprine, methotrexate, or cyclosporine) within three months prior to inclusion in the clinical trial.

Use of oral or topical probiotics within two months prior to inclusion in the clinical trial.

Use of topical or systemic antibiotics within one month prior to inclusion in the clinical trial.

Known hypersensitivity to the investigational product or any of its components.

Underlying immune-mediated diseases requiring systemic corticosteroid therapy.

Active infection in areas affected by AD requiring antibiotic, antifungal, or antiviral treatment within the one month prior to inclusion in the clinical trial.

Fever at the start of treatment (axillary temperature >37.5 °C or equivalent).

Diagnosed immunodeficiency disorders.

Current or past diagnosis of malignant neoplasms.

Any concurrent dermatologic or medical condition that, in the investigator's opinion, could interfere with the subject's response to treatment or require continuous use of topical corticosteroids.

Participation in other clinical research studies involving investigational products within one month prior to inclusion in the clinical trial.

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-11-17 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change in SCORing Atopic Dermatitis (SCORAD) after 8 weeks | 8 weeks
  Change in SCORing Atopic Dermatitis (SCORAD) index from baseline after 8 weeks of treatment with the topical emollient formulation containing Lactobacillus reuteri

SECONDARY OUTCOMES:
Change in SCORing Atopic Dermatitis (SCORAD) after 1 week | 1 week
  Change in SCORing Atopic Dermatitis (SCORAD) index from baseline after 1 week of treatment with the topical emollient formulation containing Lactobacillus reuteri
Change in SCORing Atopic Dermatitis (SCORAD) after 4 weeks | 4 weeks
  Change in SCORing Atopic Dermatitis (SCORAD) index from baseline after 4 weeks of treatment with the topical emollient formulation containing Lactobacillus reuteri
Change in POEM | 1, 4 and 8 weeks
  Change in POEM score from baseline after 1, 4, and 8 weeks of treatment with the topical emollient formulation containing Lactobacillus reuteri
Change in PIQoL-AD | 8 weeks
  Change in PIQoL-AD score from baseline after 8 weeks of treatment with the topical emollient formulation containing Lactobacillus reuteri

OTHER OUTCOMES:
Microbiota composition | Baseline and 8 weeks
  Comparative analysis of alpha and beta diversity and overall composition of the skin microbiota using high throughput 16S rRNA gene sequencing on skin swabs collected at baseline and at the end of the study.
Microbiota composition | Baseline and 8 weeks
  Comparative analysis of total bacterial load and Staphylococcus aureus load by qPCR on skin swabs collected at baseline and at the end of the study.
Adverse Events | 8 weeks
  Incidence and severity of all adverse events.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Belaneve Clinics, Alicante
  - Centro Dermatológico Estético Alicante, Alicante